CLINICAL TRIAL: NCT07211009
Title: A Single-Center, Randomized, Controlled, Phase III Clinical Study of Patient-Reported Outcome-Based Symptom Management Versus Conventional Management in Postoperative Esophageal Cancer Patients
Brief Title: Patient-Reported Symptom Care Versus Usual Care After Esophageal Cancer Surgery: A Single-Center Phase 3 Randomized Trial
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Zhen-Yu Ding, Professor, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ESO-PROSM
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Cancer (EsC)
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRO Symptom Management Group (Experimental): In the PRO arm, participants receive postoperative, PRO-based symptom management: when any target symptom score in the self-report system reaches or exceeds the predefined intervention threshold (≥2 points, indicating moderate to very severe), the system sends a real-time alert to the surgeon. The surgeon implements an intervention within the specified time window according to symptom severity. After discharge, follow-up and management are conducted via WeChat, text message, or telephone. All interventions are formulated based on relevant literature, guidelines, and expert consensus.
  Interventions: Other: Patient-Reported Outcome (PRO)-Based Symptom Management
- Conventional Management Group (Active Comparator): In the control arm, participants receive conventional postoperative symptom management. The electronic questionnaires use the same content and time points as the intervention arm, but reported symptoms do not trigger alerts, and surgeons cannot view the scores. During hospitalization, surgeons typically assess symptom severity based on patient reports during morning and afternoon rounds and manage care according to the same guidelines and consensus as the intervention arm. After discharge, no proactive symptom management is provided unless the patient actively seeks medical assistance.
  Interventions: Other: Conventional Management

INTERVENTIONS:
Other: Patient-Reported Outcome (PRO)-Based Symptom Management — Postoperative esophageal cancer patients will receive a PRO (patient-reported outcome) symptom self-report system via a WeChat mini-program/electronic form. The system covers 12 target symptoms-pain, fever, cough with sputum, dyspnea, palpitations, fatigue and activity limitation, nausea/vomiting, acid reflux/heartburn, abdominal bloating, diarrhea, swallowing obstruction (dysphagia), and hoarseness with coughing when drinking-and uses a five-level severity scale: 0 (none), 1 (mild), 2 (moderate), 3 (severe), and 4 (very severe). If any of the 12 symptom scores entered in the mini-program reaches the predefined intervention threshold (≥2, indicating moderate to very severe), the system sends a real-time alert to the surgeon, who is required to respond within a specified time window. After discharge, interventions are delivered via WeChat, text message, or telephone. Interventions mainly include counseling, patient education, prescription medication.
  Arms: PRO Symptom Management Group
Other: Conventional Management — Patients in the control arm receive conventional postoperative symptom management. The electronic questionnaires use the same content and time points as the intervention arm, but reported symptoms do not trigger alerts, and surgeons cannot view the symptom scores. During the postoperative inpatient stay, surgeons typically assess symptom severity based on patient reports during morning and afternoon rounds and manage symptoms according to the same guidelines and consensus as the intervention arm. After discharge, patients do not receive proactive symptom management from their primary surgeon unless they actively seek medical care.
  Arms: Conventional Management Group

SUMMARY:
Symptom management is fundamental to clinical care, and symptom monitoring is an effective means to detect potential adverse events early and prevent serious complications. Extensive studies show that symptom management based on patient-reported outcomes (PROs) can reduce symptom burden, improve functional status and quality of life, lower emergency visits and readmissions, and even prolong survival. However, in the field of esophageal cancer surgery, prospective clinical studies assessing the feasibility of postoperative PRO-based symptom management remain lacking. This project proposes a randomized controlled trial (RCT) in China to systematically evaluate the effectiveness and feasibility of PRO-based symptom management after esophageal cancer surgery. Through this clinical study, we aim to assess both the impact and the implementability of introducing a proactive, patient-centered PRO symptom-management model into esophageal surgical care.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years.
2. Pathologically confirmed esophageal cancer.
3. Planned to undergo curative (radical) surgical resection.
4. R0 resection.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1.
6. Adequate function of major organs.
7. Willing to complete questionnaire surveys.
8. Voluntarily agrees to participate and signs the informed consent form.
9. Good compliance and able to complete follow-up as scheduled.

Exclusion Criteria:

1. Human immunodeficiency virus (HIV) infection.
2. Psychiatric disorder.
3. Any other malignancy within the past 5 years (except completely cured carcinoma in situ of the cervix or basal cell/squamous cell carcinoma of the skin).
4. Patient ultimately did not undergo curative (radical) surgical resection.
5. Any unstable systemic disease (including active, uncontrolled gastrointestinal ulcer; active infection; grade 4 hypertension; unstable angina; congestive heart failure; unstable cerebrovascular disease; thrombotic disease; hepatic, renal, or metabolic disease; or unhealed fracture/wound as determined by the surgeon).
6. Difficulty in communication or inability to comply with long-term follow-up.
7. Any other condition deemed unsuitable by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
90-Day Postoperative Complication Rate After Esophagectomy | Postoperative days 7, 14, 30, 60, and 90, complications will be assessed and recorded at each time point.
  Proportion of patients who develop any surgery-related complication within 90 days after esophagectomy for esophageal cancer. Complication types and grades will follow the 2023 Chinese Expert Consensus on the Definition and Grading of Perioperative Complications in Esophageal and Esophagogastric Junction Cancer; complications are graded I-V, with higher grades indicating greater severity.

SECONDARY OUTCOMES:
90-Day Postoperative Mortality | Postoperative days 30, 60, and 90, death events will be recorded, and causes of death will be analyzed.
  Postoperative mortality, including death from any cause.
Number of Symptom-Threshold Events | Assess each patient-reported symptom on the day of discharge and 1 day before discharge, and on postoperative days 30, 60, and 90, and record the score for each symptom.
  Number of events in which any of the 12 target symptoms has a score ≥2.